CLINICAL TRIAL: NCT03074851
Title: Activating Mass Media for Salt Reduction Program by Using Media Reporters as Research Investigators in a Randomized Controlled Trial
Brief Title: Activating Media for Salt Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CoESeedGrant_04; CoESeedGrant_MediaReportor (Other Grant/Funding Number: united health group)
Record Dates: First submitted 2013-10-31; First posted 2017-03-09 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Hypertensive Disease
Keywords: low sodium salt; blood pressure; reporter
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salt Substitute (Experimental): To seek the relationship between blood pressure and low sodium salt.
  Interventions: Dietary Supplement: low sodium salt
- informational intervention (Other): to give 1 month informational intervention
  Interventions: Other: informational intervention

INTERVENTIONS:
Dietary Supplement: low sodium salt — To give free low sodium salt intervention for 2 months
  Arms: Salt Substitute
Other: informational intervention — to give reporter informational intervention.
  Arms: informational intervention

SUMMARY:
Mass media plays more and more important role in health education, especially in some chronic diseases which related closely with the behavior and habits. Past experience tells us that with the help of related health education in mass media such as newspaper articles, advertisements and videos on television, peoples can change their behaviors and habits in a short period of time. But when these educational information were stopped, peoples usually return to their original habits. Besides the national policy of the country how to improve the long-term health education in the mass media should be considered.This study hopes to seek an effective method to keep the mass media long-term focus on health education.

DETAILED DESCRIPTION:
In this study, reporters just like researchers were in charge of the low-sodium salt intervention. Reporters are responsible for recommended objects and measure their blood pressure personally. By observing personally the change of blood pressure pre and post low-sodium salt intervention, reporters will increase their confidence and come to the conclusion that the low salt diet is an economical way to reduce blood pressure. Those reporters would share their experiment with other people including their colleagues, Hopefully, those reporters that took part in the trial would consciously keep a sustained focus to this topic, thereby retaining a long-time education in mass media.There were two interventions. One is low-sodium salt intervention and the other is informational intervention. Low-sodium salt intervention was carried out on those family members recommended by reporters, and informational intervention. Low-sodium salt intervention was only on the reporters. The evaluation criteria of low-sodium salt intervention is the blood pressure value, and the evaluation criteria of informational intervention are the numbers of related articles in certain newspaper and the awareness of related knowledges in local population.

ELIGIBILITY:
Inclusion Criteria:

* Come from local only Daily company;
* With a national press card;
* Health Column reporters preferred;
* Without leaving plan in the next 12 months;
* With easy access to at least 4 families, including relatives, friends or neighbour;
* Volunteered to participate.

Exclusion Criteria:

* n/a

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of local media reports on salt and health | 5 years
Mean blood pressure | 2 months
  This outcome is only for the build-in randomised trial on salt substitute and blood pressure among reporters' families

SECONDARY OUTCOMES:
Awareness of knowledge on salt and health | 5 years
  A questionnaire will be applied to count the number of participants known the pre-specified answers to the questions raised on salt and health

CONTACTS AND LOCATIONS:
Overall Officials: xiangxian feng, MD, Study Director — Changzhi Medical College
Locations (1):
- Changzhi medical college, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided